CLINICAL TRIAL: NCT02435485
Title: The Rehabilitation Outcome of Patients With Lumbar Spondylolisthesis. A Prospective Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Mei-Yun Liaw, Department of physical medicine and rehabilitation, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMRPG8D0911
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Spinal Instability
Keywords: degerative lumbar spondylolisthesis; rehabilitation; balance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- spondylolisthesis with balance training (Experimental): Intervention: 1. Biodex balance training including weight shift training and random control training, 2. Regular rehabilitation including core spinal stabilization exercise.
  Interventions: Device: Biodex balance training; Other: Rehabilitation including core spinal stabilization exercise
- spondylolisthesis, no balance training (Active Comparator): Intervention: Regular rehabilitation including core spinal stabilization exercise
  Interventions: Other: Rehabilitation including core spinal stabilization exercise
- lumbar spondylitis (Active Comparator): Intervention: Regular rehabilitation including core spinal stabilization exercise
  Interventions: Other: Rehabilitation including core spinal stabilization exercise

INTERVENTIONS:
Device: Biodex balance training — 1.weight shift training, 2. random control training with Biodex balance system.
  Arms: spondylolisthesis with balance training
Other: Rehabilitation including core spinal stabilization exercise — Rehabilitation: 2-3 times a week, up to 8 weeks, 15 sessions in total. Each session will include hot packing, interferential therapy, core spine stablilzation exercise and low extremity strengthening exercise.

SUMMARY:
Patients with degenerative lumbar spondylolisthesis usually are present with low back pain, muscle spasm and weakness, radicular symptoms, intermittent claudication, insomnia, even urine or stool incontinence. There are very few research on the effectiveness of core spine stabilization exercise, balance training, and the balance effect while wearing lumbar corset in these patients.

Purpose: To investigate 1) the correlation of dynamic balance and the degree of disability with the characteristics of spinopelvic alignment. 2) potential predictors of dynamic spino-pelvic instability, 3) the effectiveness of core spine stabilization exercise, balance training and balance effect of the wearing of lumbar corset in patients with degenerative lumbar spondylolisthesis .

DETAILED DESCRIPTION:
Subjects :Seventy patients with lumbar spondylolisthesis will be randomly assigned to the group treated with balance training and without balance training, and another thirty-five age-matched lumbar spondylitis without spondylolisthesis will be assigned as control group.

Method: Patients older than 50 years of age with lumbar spondylitis or degenerative lumbar spondylolisthesis, diagnosed by KUB and lateral radiography of the lumbar-sacral spine in neutral, flexion-extension, will be recruited. Among them, seventy patients with degenerative lumbar spondylolisthesis will be recruited as experimental group and thirty-five patients with lumbar spondylitis will be recruited as control group. Exclusion criteria are patient older than 80 years of age, with stroke, spinal cord injury, head injury or other neurological deficits, previous operation of vertebrae fracture, pelvis or lower limb, isthmic lumbar spondylolisthesis, or cognitive impairment.

All subjects will receive Visual Analogue Scale (VAS), Oswestry Disability Index, Quebec back pain disability scale, and the postural stability test, 75% limits of stability test, modified clinical test of sensory integration, and the evaluation of fall risk test of Biodex balance system at beginning and at the end of program. Both the control and experimental groups will receive rehabilitation training, including hot packing, interferential therapy, core spine stabilization exercise and lower extremity strengthening exercise for 2-3 times a week, up to 8 weeks, 15 sessions in total. Patients in the experimental group will be randomly assigned to either a balance training group or to a group without balance training. The balance training will include both weight shift training and random control training with Biodex balance system. A balance effect of wearing lumbar corset will be evaluated at the beginning of the program. The investigators will follow up with these patients by telephone 3 months after program completion.

The clinical history, age, gender, body weight, body height, job, symptoms and sign, Visual Analogue Scalce (VAS), Questionnairem (Quebec back pain disability scale) and Oswestry Disability Index will be recorded at base and after rehabilitation program. Every subject will sign the informed consent, which will be obtained from the Institutional Review Board of Chang Gung Memorial Hospital.

Physical examination It will include the duration, pain intensity, neurologic deficits, muscle power of lower limbs, deep tendon reflex, sensation, stretch sign or nerve conduction velocity, or electromyography examination.

Radiography All subjects will receive Kidney Ureter Bladder (KUB) and standing lateral radiography of lumbar-sacral spine in neutral, to determine the pelvic incidence, pelvic tilt, sacral slope etc. Furthermore the patients with spondylolisthesis will receive flexion-extension of lumbar-sacral spine to determine the degree of translational motion of vertebrae.

Rehabilitation Correct body posture and lifting techniques will be instructed. After patient's back pain subside to a degree of less than 5 of visual analogue scale (VAS), balance test will be assessed by using the Biodex Balance System (BBS), including postual stability test, limits of stability test, modified clinical test of sensory intergration and fall risk test. The spondylolisthesis patients will be assessed while wearing or without wearing lumbar corset at the beginning of the program, which will be tested in a random order. The tester for BBS will be blind to the patient's grouping. The anterio-posterior, medial-lateral stability index and overall stability index etc will be recorded.

Both groups will receive 2-3 times a week, up to 8 weeks, 15 sessions in total. Each session will include 15-minute hot packing, 15-minutes interferential therapy, about 25 minutes of core spine stablilzation exercise and low extremity strengthening exercise on the stationary bicycle. And patients in the experimental group will be randomly assigned either to a balance training group or to a group without balance training. The balance training will include both weight shift training and random control training with Biodex balance system. A balance effect of wearing lumbar corset will be evaluated at the beginning of the program.

Balance test

1. Postual stability test: Patients will stand barefoot on the platform with a slight knee flexion, look straight ahead with arms across the chest on the platform, and then subject will be asked to maintain a quiet stance on the platform for seconds for initialization. Six stability trials will be performed with eyes open and eyes closed over a period of 20 seconds, 3 trials per each state, with 10-second count rest countdown in between the trials.
2. Limits of stabitiy (LOS) test (75% LOS): an indicator of dynamic control within a normalized envelope. Nine targets blink in random order on the screen. Patient have to shift body weight to move the cursor frorm the center target to a blinking target and back as quickly and with as little deviation as possible. The overall direction control of overall, forward, backward, right, left, forward/right, forward/right, backward/right and backward/left will be recorded.
3. Modified clinical test of sensory intergration: It consists of the first condition: eye open with firm surface, the second condition: eye closed with firm surface, the third condition: eye open with foam surface and the fourth condition: eye closed with foam surface
4. Fall risk test: to identify the high potential fall risk patient.

Rehabilitation program (Home base or outpatient training) Education: Both of home base and outpatient training patients will be instructed to use superficial heat for relief of back pain, muscle spasm; and correct posture of the activities of daily living (sitting, standing, sleeping, working and driving), lifting techniques, avoidance of certain movements and postures, such as prolonged standing or sitting, slouched in a soft armchair, sagging bed mattresses, wearing high heels or carrying heavy objects. And lumbar corset for stabilization of spine will be recommended.

Outpatient program: Two to three times a week, 15 treatment sessions, about 60 minutes per session, up to 8 weeks. It will include hot pack and/or interferential therapy about 15 minutes. Exercise (about 25 min) will begin with a short warm-up aerobic exercise, upper back and shoulder extension exercise, pectoral stretching exercise, back extension exercise, combined with deep-breathing exercise; then a core strengthening program, including cat and camel, abdominal hollowing, bridge, dead bug, quadruped etc. The exercise will be 3 sessions of 10-15 repetitions.

Balance training Balance training: same as rehabilitation program (total 15 sessions, 2-3 times a weeks)

1. Weight shifting training Guiding moving point (a) from quarter one to quarter three, (b) from quarter two to quarter four, (c) in parallel to the vertical line in the feedback screen (anterior-posterior direction)
2. Random training It is ideal for motor control and vestibular training. Static mode : work within the sway envelope to move the cursor and attempt to keep it within the moving target.

Dynamic mode: use hip, knee and ankle strategies to manipulate the moving palteform's cursor to within the random moving target.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 50 years of age with lumbar spondylitis or degenerative lumbar spondylolisthesis, low back pain, or radicular symptoms and diagnosed by KUB and lateral radiography of the lumbar-sacral spine in neutral, flexion-extension, will be recruited. Among them, seventy patients with degenerative lumbar spondylolisthesis as the experimental group and thirty-five patients with lumbar spondylitis will be included as the control group.

Exclusion Criteria:

* Patient older than 80 years of age, with stroke, spinal cord injury, head injury or other neurological deficits, previous operation of vertebrae fracture, pelvis or lower limb, isthmic lumbar spondylolisthesis, or cognitive impairment. -

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Biodex balance test | 8 weeks, 6 months
  1. Postural stability test: overall index___, anterior-posterior index___, medial-lateral index____
  2. Limits of stability test: forward___, backward___, right___, left___, forward/right___, forward/left___, backward/right___, backward/left___
  3. Modified clinical test of sensory integration: sway index: eye open, firm___; eye close,firm___, eye open, foam___, eye close foam___
  4. Fall risk test: actual score, STD_______

SECONDARY OUTCOMES:
Oswestry Disability Index (Oswestry Low Back Pain Disability Questionnaire) | 8 week, 6 months
  To measure a patient's permanent functional disability
Quebec back pain disability scale | 8 weeks, 6 months
  This questionnaire is about the way patient's back pain affecting their daily life
Visual analog scale (VAS) of low back pain and radicular pain | 8 weeks, 6 months
  Visual analog scale [VAS] is a measure of pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Yun Liaw, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Kaohsiung Chang Gung Memorial Hospital.
Locations (1):
- Department of Physical Medicine and Rehabilitation, Kaohsiung Chang Gung Memorial Hospital., Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No